CLINICAL TRIAL: NCT02935101
Title: Effects of Glucocorticoids on Craving During Detoxification Treatment of Heroin and/or Stimulants
Acronym: Goliath
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulties in recruiting study participants
Sponsor: Prof. Dominique de Quervain, MD (Other)
Collaborators: Psychiatric Hospital of the University of Basel (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, Director Division Cognitive Neuroscience, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2016-00851
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Opioid Dependence; Cocaine Dependence
Keywords: glucocorticoids; craving; Heroin; Cocaine; dependency
MeSH Terms: conditions — Opioid-Related Disorders; Cocaine-Related Disorders | interventions — Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prednisolon (Experimental): Participants will receive an oral administration of prednisolone or placebo two times daily for the first five days of opioid detoxification, starting after one day of regular detoxification as baseline. Oral prednisolone will be administered in a dose consistent with standard treatment guidelines for glucocorticoid deficiency (Oelkers, 1996).
  Interventions: Drug: Prednisolone
- Placebo (Placebo Comparator): Identical looking capsules like the IMP containing placebo (without active component) for oral administration.
  Interventions: Drug: Placebo (for Prednisolone)

INTERVENTIONS:
Drug: Prednisolone — formulated for oral administration. encapsulated.
  Other Names: Prednisolon Streuli(R)
  Arms: Prednisolon
Drug: Placebo (for Prednisolone) — Sugar pill manufactured to mimic Prednisolon 10mg capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate whether prednisolone lowers intensity and frequency of craving in heroin-addicted subjects undertaking a detoxification of cocaine and/or heroin.

DETAILED DESCRIPTION:
Participants of this study are 120 heroin-addicted patients who are inward for a detoxification program for either cocaine or cocaine and heroin. Depending on the detoxification substance(s) there will be two groups of participants: Detoxification of cocaine (A; 60 participants) and detoxification of heroin and cocaine (B; 60 participants). The detoxification starts mandatory with the admission to the ward and lasts about 1-2 weeks. The participation in the study lasts about 4-5 weeks (including follow-up visits). Intake of study medication starts two days after admission and one day after informed consent. Each participant will get either 30mg/d prednisolon or placebo during five days. Participants will be under normal medical supervision during the treatment phase until follow-up 2 (final examination) provided by ward staff. Treatment days and follow-up 1 and 2 consist of : (1) vital signs (BP, HR, temperature) as measured in the daily routine, (2) at midday: visual analogue scales asking about craving for heroin and cocaine at the moment, (3) afternoon: questionnaires to survey mainly the withdrawal symptoms and vegetative parameters.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature,
* age ≥18,

  * Group A Detoxification of stimulants (cocaine, amphetamine and/or methamphetamine); ICD-10: F14.2 and/or F15.2) OR Stable opioid dependency (no parallel consumption). Detoxifica-tion of stimulants.
  * Group B Opioid dependency and dependency of stimulants (cocaine, amphetamine and/or methamphetamine) and Detoxification of parallel consumption of stimulants and heroin (ICD-10: F11.2, 14.2, 15.2)
* admission for detoxification to ward U2 of the University Psychiatric Hospital of Basel

Exclusion Criteria:

* contraindications to the class of drugs under study or to any of the excipients, e.g. known hypersensitivity or allergy to class of drugs or the investigational product;
* acute or severe co-morbid psychiatric disturbances (such as a heavy episode of major depression with suicidal ideations, acute exacerbation of a bipolar disorder, acute exacerbation of schizophrenia, alcohol addiction with an acute relapse, psychosis, dementia);
* current medical conditions excluding participation (such as acute infectious disease, moni-tored by elevated CRP, diabetes mellitus, anticoagulation therapy);
* recent history of systemic or topic glucocorticoid therapy;
* alcohol intake > 0.0 ‰ according to breathalyser test on day 0 (screening) to exclude severe alcohol abuse;
* specific drugs not allowed during the study or for specific periods of time prior to the administration of the test dose: Anticoagulant agents, antidiabetic agents, cyclosporine;
* women who are pregnant or breast feeding;
* intention to become pregnant during the course of the study;
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia;
* participation in another study with investigational drug within the 30 days preceding or during the present study;
* previous enrolment into the current study;
* enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Heroin Craving | Assessing change between baseline and some predefined time points during 2 weeks
  Heroin Craving Questionnaire, 14 items (HCQ; Tiffany et al., 1993 and Heinz et al., 2006)
Cocaine Craving | Assessing change between baseline and some predefined time points during 2 weeks
  Cocaine Craving Questionnaire, 14 items (CCQ; Tiffany et al., 1993 and Heinz et al., 2006)
Heroin Craving | Assessing change between baseline and some predefined time points during 2 weeks
  Visual Analogue Scale Craving
Cocaine Craving | Assessing change between baseline and some predefined time points during 2 weeks
  Visual Analogue Scale Craving

SECONDARY OUTCOMES:
Withdrawal Symptoms according to ICD-10 (F14.3 and F12.2) | Assessing change between baseline and some predefined time points during 2 weeks
Questionnaire 'Health State' | Assessing change between baseline and some predefined time points during 2 weeks
  SF-12 (Morfeld M. et al., 2011)
Questionnaire 'Anger/Irritation' | Assessing change between baseline and some predefined time points during 2 weeks
  STAI-G form X1 (state; Laux L. et al., 1981)
Questionnaire 'Anxiety' | Assessing change between baseline and some predefined time points during 2 weeks
  STAXI (Schwenkmezger P. et al., 1992/2006)
Saliva Cortisol levels | Assessing change between baseline and some predefined time points during 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Antje Kemter, MD, Principal Investigator — UPK Basel
Locations (1):
- Psychiatric Hospital University of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided